CLINICAL TRIAL: NCT04710316
Title: Étude de l'épidémie de SARS-CoV-2 Dans Les Services Hospitaliers de Bamako, Mali
Brief Title: Study of COVID-19 Outbreak in Hospital Departments of Bamako, Mali
Acronym: BAMACOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C20-41
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-01

CONDITIONS: Covid19
Keywords: Covid-19; SARS-CoV-2; Mali; Africa; Hospital
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Interventions
  * Serological screening of caregivers at D0, M1, M2, M3.
  * Screening of patients by molecular biology: a nasopharyngeal swab will be performed to symptomatic hospitalized patients or who have been in close contact with a SARS-CoV-2 infected person without effective protective measures to search for SARS-CoV-2 genome. Positive clinical isolates will be sequenced.
  * Screening of caregivers by molecular biology: a nasopharyngeal swab will be performed to symptomatic caregivers or who have seroconverted to SARS-CoV-2 or who have been in close contact with a SARS-CoV-2 infected person without effective protective measures to search for SARS-CoV-2 genome. Positive clinical isolates will be sequenced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): - Hospitalized patients in one of the four centers in Bamako, with clinical signs of infection of the upper or lower respiratory tracts with fever or feeling of fever or any other signs of SARS-Cov-2 infection or who have been in close contact with a SARS-CoV-2 infected person without effective protective measures
  Interventions: Diagnostic Test: SARS-CoV-2 screening by molecular biology
- Caregivers (Experimental): Caregivers of one of the four centers in Bamako.
  * Serological screening: all.
  * Molecular screening: with clinical signs of infection of the upper or lower respiratory tracts with fever or feeling of fever or any other signs of SARS-Cov-2 infection or who have seroconverted to SARS-CoV-2 or who have been in close contact with a SARS-CoV-2 infected person without effective protective measures
  Interventions: Diagnostic Test: SARS-CoV-2 screening by molecular biology; Diagnostic Test: Serological screening

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 screening by molecular biology — SARS-CoV-2 RT-PCR in nasopharyngeal swab targeting 2 regions of the viral genome
Diagnostic Test: Serological screening — Serological screening of caregivers at D0, M1, M2, M3 (anti-nucleocapsid antibodies).
  Arms: Caregivers

SUMMARY:
The new coronavirus known as SARS-Cov-2 (severe acute respiratory syndrome -coronavirus 2) was first reported in December 2019 and rapidly became a public health emergency. The COVID-19 pandemic is now affecting sensitive regions with fragile health care systems, such as South America and Africa. Caregivers, in the front line of Covid19 patient management, may accidentally become infected and a source of infection during the incubation phase or in case of asymptomatic infection.

The objectives of this project are thus i) to assess SARS-Cov-2 spread over the hospital departments of Bamako by carrying out a systematic molecular screening of patients and caregivers, ii) to evaluate the feasibility of Point-Of-Care molecular assays in Mali and iii) to estimate the immunity acquired from SARS-Cov-2 among health workers through serological testing, allowing also the assessment of asymptomatic caregiver rate and absence of re-infection among the immunized caregivers. Finally, iv) variability of the virus over time and spread of different variants around the world will be studied by sequencing the viral genome.

ELIGIBILITY:
Inclusion Criteria:

* Free and informed consent accepted in writing
* Patient: patient hospitalized in one of the four hospitals of Bamako, with clinical signs of infection of the upper or lower respiratory tracts (sore throat, cough/sputum, nasal congestion and rhinorrhea, odynophagia, thoracic oppression, dyspnea, desaturation) with fever or feeling of fever or any other signs of SARS-Cov-2 infection (that is to say the following clinical manifestations, of sudden onset: unexplained asthenia, unexplained myalgia, headache without a known migraine disease, anosmia or hyposmia without associated rhinitis, dysgueusia, diarrhea, heart rhythm disorders, acute myocardial injury, severe thromboembolic event) or who have been in close contact with a SARS-CoV-2 infected person without effective protective measures (FFP2/surgical masks or physical separation) and defined as follows: having shared the same place of life as the confirmed case, for example: family, same room or having a direct contact in face to face with less than 1 meter from the confirmed case during a talk; intimate friends; class or office neighbours; adjacent to the index case in a plane or a train; or having provided or received hygiene or care acts from a confirmed case.
* Caregivers: caregivers of one of the four hospitals of Bamako

Exclusion Criteria:

* Persons subject to legal protection or not able to give a free and informed consent.
* Caregivers: caregivers not able to follow the project schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence rate of positive SARS-Cov-2 RT-PCR in Bamako hospital departments during the study | Through the completion of subject participation (up to 15 months after study start date).
  Positive SARS-Cov-2 RT-PCRs are defined by the detection of SARS-Cov-2 genome after amplification using a test targeting 2 regions of the genome.

SECONDARY OUTCOMES:
Number of Cepheid Xpert® Xpress SARS-Cov-2 cartridges available for 19.8 USD/number required for the project | Through the completion of subject participation (up to 15 months after study start date).
Percentage of positive serological tests among the caregivers of the hospital departments of Bamako. | Assessed on the fourth serological assay performed (at Month 3).
Percentage of caregivers asymptomatic but immunized to SARS-CoV-2 | Assessed on the fourth serological assay performed (at Month 3).
Percentage of caregivers immunized and re-infected with SARS-CoV-2 | Through the completion of caregiver participation (up to 15 months after study start date).
Number of SARS-CoV-2 mutations/variants detected during the study | Through the completion of subject participation (up to 15 months after study start date).
Percentage of SARS-CoV-2 mutations/variants detected during the study | Through the completion of subject participation (up to 15 months after study start date).

CONTACTS AND LOCATIONS:
Overall Officials: Almoustapha Issiaka MAIGA, Principal Investigator — SEREFO/UCRC, FMOS - University Hospital Gabriel Toure, Bamako, Mali; Eve Todesco, Principal Investigator — APHP - Sorbonne university
Locations (4):
- Mali (4):
  - Hopital du Point-G, Bamako
  - Hopital Gabriel Toure, Bamako
  - Hôpital dermatologique de Bamako, Bamako
  - Hôpital du Mali, Bamako

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maiga AI, Saliou M, Kodio A, Traore AM, Dabo G, Flandre P, Fofana DB, Ammour K, Tra NOME, Dolo O, Marcelin AG, Todesco E. High SARS-CoV-2 seroprevalence among health care workers in Bamako referral hospitals: a prospective multisite cross-sectional study (ANRS COV11). Clin Microbiol Infect. 2022 Jun;28(6):900-902. doi: 10.1016/j.cmi.2022.02.019. Epub 2022 Feb 16. No abstract available. PMID 35182761